CLINICAL TRIAL: NCT01264536
Title: Pilot Study: Lactoferrin for Prevention of Neonatal Sepsis
Acronym: NEOLACTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Theresa Ochoa, Assistant Professor of Pediatrics, Universidad Peruana Cayetano Heredia, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIDISI 56909; OPP1015669 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Sepsis
Keywords: lactoferrin; sepsis; neonates; prevention; infections
MeSH Terms: conditions — Sepsis; Infections | interventions — Lactoferrin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactoferrin (Experimental): Lactoferrin is a freeze-dried protein purified directly from fresh bovine milk.
  Interventions: Dietary Supplement: lactoferrin
- maltodextrin (Placebo Comparator): Maltodextrin is an inert sugar.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: lactoferrin — Infants will receive oral bovine lactoferrin (200 mg/Kg/day divided in three dosis) for 4 weeks. Lactoferrin will be dissolved in human milk or infant formula or in a 5% glucose solution. Each dose will be dissolved in a small volume so the maximum lactoferrin concentration will be 25mg/mL.
  Other Names: Bovine lactoferrin
  Arms: Lactoferrin
Dietary Supplement: Maltodextrin — Infants will receive oral maltodextrin (200mg/Kg/day in three divided dosis) for 4 weeks. Maltodextrin will be dissolved in human milk or infant formula or in a 5% glucose solution. Each dose will be dissolved in a small volume so the maximum maltodextrin concentration will be 25mg/mL.
  Arms: maltodextrin

SUMMARY:
We will test the hypothesis that bovine lactoferrin supplementation prevents serious infections in preterm infants. We will conduct a randomized placebo-controlled double blind study in 190 premature infants <2500 gm in 5 Neonatal Intermediate and Intensive Care Units in Lima, Peru to determine whether bovine lactoferrin prevents the first episode of late-onset sepsis.

DETAILED DESCRIPTION:
Lactoferrin is an iron chelating protein with multiple physiological functions (anti-microbial, anti-inflammatory and immunomodulatory) and is one of the most important proteins present in mammalian milk. We hypothesize that lactoferrin as an oral supplement given daily to low birth weight will improve their health by mimicking their protective role in milk. There is extensive literature showing in vitro and in animal models the benefits of lactoferrin. However, there are few clinical trials designed to translate this knowledge into patient care.

We will conduct a pilot randomized, double-blinded placebo-controlled trial comparing daily supplementation with bovine lactoferrin versus placebo in neonates to reduce the incidence of sepsis in the first month of life. We will enroll 190 neonates with a birth weight less than 2,500 g, younger than 3 days of age in the neonatal intensive care unit of 5 pediatric hospitals in Lima, after informed consent of both parents. Infants will be followed in the hospital until death or discharge and then at home up to 1 month of age. Bovine lactoferrin will be used in this trial (200 mg/Kg per day). Although bovine and human lactoferrin are not identical, their bioactivity is quite comparable. Maltodextrin (an inert sugar) will be used for controls. The primary study outcome will be the number of first late-onset sepsis episodes (occurring >72h after birth with isolation of any pathogen in blood or cerebrospinal fluid).

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with a birth weight between 500g and 2500g
2. Neonates born in, or referred to the Neonatal Intermediate and Intensive Care Units of one of the participating hospitals in the first 72 hours of life.

Exclusion Criteria:

1. Neonates with underlying gastrointestinal problems that prevent oral intake.
2. Neonates with predisposing conditions that profoundly affect growth and development (chromosomal abnormalities, structural brain anomalies, severe congenital abnormalities)
3. Neonates with a family background of cow milk allergy
4. Neonates that, according to the investigator criteria, will not have the chance to complete the subsequent study visits (patients that before one month old would not be living in Lima).
5. Neonates whose parents decline to participate.

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of confirmed episodes of late-onset sepsis. | 1 month
  Number of confirmed episodes of late-onset sepsis in the first month of life

SECONDARY OUTCOMES:
Incidence of Gram positive and Gram negative bacterial and fungal bouts of sepsis, pneumonia, diarrhea and mortality | 1 month
  Incidence of Gram positive and Gram negative bacterial and fungal bouts of sepsis, pneumonia, diarrhea and mortality in the first month of life.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa J Ochoa, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (3):
- Peru (3):
  - Hospital Guillermo Almnara Irigoyen, Lima, Lima Province
  - Hospital Nacional Cayetano Heredia, Lima, Lima Province
  - Hospital Nacional Alberto Sabogal Sologuren, Callao, Lima

REFERENCES:
- [Background] Manzoni P, Rinaldi M, Cattani S, Pugni L, Romeo MG, Messner H, Stolfi I, Decembrino L, Laforgia N, Vagnarelli F, Memo L, Bordignon L, Saia OS, Maule M, Gallo E, Mostert M, Magnani C, Quercia M, Bollani L, Pedicino R, Renzullo L, Betta P, Mosca F, Ferrari F, Magaldi R, Stronati M, Farina D; Italian Task Force for the Study and Prevention of Neonatal Fungal Infections, Italian Society of Neonatology. Bovine lactoferrin supplementation for prevention of late-onset sepsis in very low-birth-weight neonates: a randomized trial. JAMA. 2009 Oct 7;302(13):1421-8. doi: 10.1001/jama.2009.1403. PMID 19809023
- [Derived] Ochoa TJ, Zegarra J, Cam L, Llanos R, Pezo A, Cruz K, Zea-Vera A, Carcamo C, Campos M, Bellomo S; NEOLACTO Research Group. Randomized controlled trial of lactoferrin for prevention of sepsis in peruvian neonates less than 2500 g. Pediatr Infect Dis J. 2015 Jun;34(6):571-6. doi: 10.1097/INF.0000000000000593. PMID 25973934